CLINICAL TRIAL: NCT02871518
Title: A Randomized Phase II Non-inferiority Study of Two Cycles Versus Three Cycles of Cisplatin Based Concurrent Chemoradiotherapy for Low Risk Locoregionally Advanced Nasopharyngeal Carcinoma Based on Pretreatment Plasma EBV DNA Level
Brief Title: Two Cycles Versus Three Cyclle of CCRT for Low Risk Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, the vice director of nasopharyngeal carcinoma, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cycle of CCRT and NPC
Record Dates: First submitted 2016-07-17; First posted 2016-08-18 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Two cycle CCRT (Experimental): Concurrent cisplatin(100mg/m2,D1,D22)combine with IMRT
  Interventions: Drug: Cisplatin combine with IMRT
- Three cycle CCRT (Active Comparator): Concurrent cisplatin(100mg/m2,D1,D22 and D43)combine with IMRT
  Interventions: Drug: Cisplatin combine with IMRT

INTERVENTIONS:
Drug: Cisplatin combine with IMRT — Concurrent cisplatin (100mg/m2，D1,D22) combine with IMRT
  Other Names: DDP
  Arms: Two cycle CCRT
Drug: Cisplatin combine with IMRT — Concurrent cisplatin (100mg/m2，D1,D22 and D43) combine with IMRT
  Other Names: DDP
  Arms: Three cycle CCRT

SUMMARY:
This is a Phase II trial to study the effectiveness of two cycles versus three cycles of Concurrent Chemoradiotherapy in treating patients with Low Risk Locoregionally Advanced Nasopharyngeal Carcinoma based on pretreatment plasma EBV DNA.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is endemic in Southern China and Southeast Asia. Several prospective randomized trials have demonstrated that concurrent chemoradiotherapy was superior to radiotherapy alone in the treatment of locoregionally advanced NPC. Concurrently, although cisplatin-based concurrent chemoradiotherapy was considered as the standard regimen for locoregionally advanced nasopharyngeal carcinoma, several prospective randomized trials have demonstrated that only 52-63% patients can finished three cycles cisplatin-based concurrent chemoradiotherapy( DDP, 100mg/m2,D1,D22 and D43), due to chemoradiotherapy induced toxicity. Combined analyses of NPC-9901 and NPC-9902 Trials indicated that the 5-year locoregional failure free survival was insignificant between the patients received between two and three cycles cisplatin-based concurrent chemoradiotherapy. Our previous studies have also demonstrated that the five years overall survival, distant metastasis free survival and 5-year locoregional failure free survival was not observed significant difference between the patients received between two and three cycles cisplatin-based concurrent chemotherapy. It indicated that one pressing questions remain to be resolved: can we define the optimal dose so that we can reduce toxicity by avoiding unnecessary overdose or an ineffective phase of treatment? Recently, the quantification of pretreatment plasma Epstein-Barr virus (EBV) DNA, which was considered the most potential biomarker to compliment TNM stage, was demonstrated a useful biomarker for the risk stratification, monitoring and prediction of the prognosis of NPC. The investigators previous study demonstrated that for local and regionally advanced NPC patients with EBV DNA <4,000copies/mL, the 3-year's PFS and DMFS was approximate to 90%. Pretreatment plasma EBV DNA levels might be applied to guide concurrent chemotherapy regimen for local and regionally advanced NPC patients. Therefore, the investigators make a hypothesis that the low risk locoregionally advanced NPC patients received two cycles of chemotherapy may gain similar long-term survival as those received three cycles of chemotherapy, leading to less chemotherapy induced toxicity. Therefore, this phase II non-inferiority, randomised controlled clinical trial was designed to assess efficacy for low-risk patients, identified with pretreatment plasma EBV DNA <4,000 copies/mL, received two cycle cisplatin-based chemotherapy compared with three cycle cisplatin-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
* Original clinical staged as T3-4N0-3 M0 or any T、N2-3M0（according to the 7th AJCC edition）
* No evidence of distant metastasis (M0)
* Pretreatment Plasm EB Virus DNA<4000copies/ml
* Male and no pregnant female
* Satisfactory performance status: ECOG (Eastern Cooperative OncologyGroup) scale 0-1
* WBC ≥ 4×109 /L and PLT ≥4×109 /L and HGB ≥90 g/L
* With normal liver function test (ALT、AST ≤ 2.5×ULN, TBIL≤ 2.0×ULN)
* With normal renal function test (Creatinine ≤ 1.5×ULN)

Exclusion Criteria:

* Patients have evidence of relapse or distant metastasis
* Histologically confirmed keratinizing squamous cell carcinoma (WHO I)
* Receiving radiotherapy or chemotherapy previously
* The presence of uncontrolled life-threatening illness
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Receiving other ways of anti-cancer therapy.
* Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | 3 years
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up

SECONDARY OUTCOMES:
The shor-term toxic effects | 3 months
  The shorterm toxic effects were assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0)
Complete Response (CR) | after the completion of the chemoradiotherapy treatment (up to 9 weeks)
  CR assessed by independent reviewers, according to the Modified Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the chemoradiotherapy treatment. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) only
Overall Survival(OS) | 3 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up
Locoregional Relapse-Free Survival(LRRFS) | 3 years
  The LRRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit
Distant Metastasis-Free Survival (DMFS) | 3 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit
Cost-effectiveness analysis | 3 years
  The cost (including direct cost drug fees, inspection fees, expenses and nursing cost) and incremental cost-effectiveness ratio was calculated between two arms
The monitoring of plasma EBV DNA | 3 years
  The plasma EBV DNA will be detected before treatment ,during treatment (weekly) and during follow up( every 3-6 months)
Long-term toxicities | 3 years
  Patients will be monitored for long-term toxicity by standard NIH criteria. QoL was assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) and EORTC QLQ Head and Neck

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li YC, Li XY, Lan KQ, Cheng H, Chen J, Liu LT, Wen DX, Gu LW, Guo WP, Sun XS, Liu SL, Yang JH, Li SC, Li YF, Long HX, Luo DH, Guo L, Mo HY, Sun R, Guo SS, Wang P, Li LB, Yang Q, Liang YJ, Jia GD, Yan JJ, Zhao C, Chen QY, Li LJ, Mai HQ, Tang LQ. Epstein-Barr virus DNA-guided chemoradiotherapy for patients with low-risk locoregionally advanced nasopharyngeal carcinoma: a secondary 5-year follow-up analysis of an open-label, randomised controlled, phase 2 non-inferiority trial. EClinicalMedicine. 2025 Oct 30;90:103615. doi: 10.1016/j.eclinm.2025.103615. eCollection 2025 Dec. PMID 41245547
- [Derived] Li XY, Luo DH, Guo L, Mo HY, Sun R, Guo SS, Liu LT, Yang ZC, Yang JH, Qiu F, Sun XS, Wang P, Liu Q, Li JB, Tang QN, Lin C, Yang Q, Liu SL, Liang YJ, Jia GD, Wen DX, Guo CY, Yan JJ, Zhao C, Chen QY, Tang LQ, Mai HQ. Deintensified Chemoradiotherapy for Pretreatment Epstein-Barr Virus DNA-Selected Low-Risk Locoregionally Advanced Nasopharyngeal Carcinoma: A Phase II Randomized Noninferiority Trial. J Clin Oncol. 2022 Apr 10;40(11):1163-1173. doi: 10.1200/JCO.21.01467. Epub 2022 Jan 6. PMID 34990291